CLINICAL TRIAL: NCT01984164
Title: CAndesartan vs LIsinopril Effects on the BRain and Endothelial Function in eXecutive MCI (CALIBREX)
Brief Title: CAndesartan vs LIsinopril Effects on the BRain
Acronym: CALIBREX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Ihab Hajjar, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00070087; R01AG042127 (NIH)
Record Dates: First submitted 2013-10-27; First posted 2013-11-14 (Estimated); Results first posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Hypertension; Mild Cognitive Impairment
Keywords: Cerebrovascular function
MeSH Terms: conditions — Hypertension; Cognitive Dysfunction | interventions — candesartan; candesartan cilexetil; Lisinopril

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Candesartan (Active Comparator): To achieve blood pressure control, we will use a stepwise protocol as follows: candesartan (blinded) 8mg→ 16mg→ 32mg. Both groups will also receive (unblinded) , if needed to achieve blood pressure control, HCTZ 12.5mg→ 25mg, Amlodipine 2.5mg→ 5mg →10mg and metoprolol succinate extended release 12.5mg→ 25mg→ 50mg. Antihypertensive medications will be increased every 2 weeks until control is achieved.
  Interventions: Drug: Candesartan
- Lisinopril (Active Comparator): To achieve blood pressure control we will use a stepwise protocol as follows: lisinopril (blinded) 10mg→ 20mg→ 40mg. Both groups will also receive (unblinded), if needed to achieve blood pressure control, HCTZ 12.5mg→ 25mg, Amlodipine 2.5mg→ 5mg→ 10mg and metoprolol succinate extended release 12.5mg→ 25mg→ 50mg. Antihypertensive medications will be increased every 2 weeks until control is achieved.
  Interventions: Drug: Lisinopril

INTERVENTIONS:
Drug: Candesartan — blinded
  Other Names: Atacand
  Arms: Candesartan
Drug: Lisinopril — Blinded
  Arms: Lisinopril

SUMMARY:
The aim of this study is to conduct a 1-year double blind randomized control trial comparing candesartan to lisinopril in 140 individuals with hypertension and executive mild cognitive impairment in their effects on executive function, neuroimaging markers, and vascular indicators.

DETAILED DESCRIPTION:
* Hypertension is associated with cognitive impairment even in the absence of clinical dementia. To date, no specific treatment is available for this pattern of mild cognitive impairment related to hypertension.
* Objectives or purpose: The aims of this study are to investigate the effects of candesartan on executive function decline and on changes in cerebral perfusion, cerebrovascular reserve and microvascular brain injury. The study also intends to identify potential underlying mechanisms related to vascular structure and function, including atherosclerosis, vascular inflammation, vascular stiffness, and endothelial progenitor cells, by which candesartan may affect the cognitive and cerebrovascular outcomes.
* Study methodology:This is a double blind randomized clinical trial that will be conducted in 140 individuals (70 in the candesartan group, 70 in the lisinopril group). Our target population is subjects: 55 years or older with hypertension and Executive Mild Cognitive Impairment.
* Endpoints to be measured:Our measures include cognitive function, cerebral perfusion and reserve, markers of vascular brain damage, atherosclerosis, stiffness, vascular inflammation and endothelial function.
* Description of intervention, follow-up, and duration of study: Eligible participants will undergo randomization into 2 groups and will be seen frequently until their blood pressure is controlled (<140/90 mmHg). Participants will be seen at 3, 6 and 12 months afterwards.

ELIGIBILITY:
Inclusion Criteria:

1. age: 55 years or older;
2. Hypertension: SBP≥140 mm Hg or DBP≥ 90 mm or receiving antihypertensive medications.
3. Executive MCI will be defined using these criteria:

   1. The Montreal Cognitive Assessment (MoCA) score less than or equal to 26
   2. Executive dysfunction: A performance at the 10th percentile or below on at least one of four screening tests for executive function: Trail Making Test, Part B (TMT-B), modified Stroop interference, Digit Span and Digit Sequencing, and Letter fluency.
   3. Minimal Functional limitation as reflected by the Functional Assessment Questionnaire (FAQ)≤7

Exclusion Criteria:

1. Intolerance to study drugs;
2. SBP >200 or DBP >110 mm Hg;
3. Renal disease or hyperkalemia
4. Active medical or psychiatric problems
5. Uncontrolled congestive heart failure;
6. History of stroke in the past 3 years;
7. Inability to perform the study procedures
8. Women of childbearing potential
9. diagnosis of dementia
10. In those who lack decision capacity, a study surrogate who can sign on their behalf will be required. Since we are enrolling only those with MCI, we anticipate that most participants will have decision capacity
11. Current use of Lithium, as most antihypertensive classes may lead to increased lithium toxic levels.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2014-08-20 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2018-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ihab Hajjar, MD, MS, Principal Investigator — Emory Univeristy
Locations (1):
- Emory Univeristy, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Hajjar I, Okafor M, McDaniel D, Obideen M, Dee E, Shokouhi M, Quyyumi AA, Levey A, Goldstein F. Effects of Candesartan vs Lisinopril on Neurocognitive Function in Older Adults With Executive Mild Cognitive Impairment: A Randomized Clinical Trial. JAMA Netw Open. 2020 Aug 3;3(8):e2012252. doi: 10.1001/jamanetworkopen.2020.12252. PMID 32761160

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Candesartan | Lisinopril
Started | 87 | 89
Completed | 77 | 64
Not Completed | 10 | 25
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Adverse Event | 5 | 19
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Candesartan | Lisinopril | Total
Number analyzed (Participants) | 87 | 89 | 176
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.1 (8.3) | 65.8 (7.2) | 65.9 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 54 | 101
  Male | 40 | 35 | 75
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 56 | 57 | 113
  White | 29 | 31 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants] — Of 176 eligible participants enrolled and randomized to candesartan or lisinopril, 35 dropped out before study completion (25 from the lisinopril arm and 10 from the candesartan arm). The final sample for the intention-to-treat analysis was 141 individuals, including 77 in the candesartan group and 64 in the lisinopril group.
  participants
    United States | 87 | 89 | 176
MoCA score [Mean (Standard Deviation); unit: points] — MoCA is a 30-point scale administered in 10 minutes, is validated in Spanish and is highly sensitive to identify mild vascular-related cognitive dysfunction. MoCA includes assessment of MoCA assesses: Short term memory, visuospatial abilities, executive functions, attention, concentration and working memory, language and orientation to time and place. Scale is 0-30 with higher indicated better cognitive performance.
  points | 21.4 (3.4) | 21.7 (3.5) | 21.5 (3.4)

OUTCOME MEASURES:

1. Primary Outcome: Executive Function
Description: Executive function will be assessed using Trail Making Test (part B-A). Part A was collected to correct for motor speed and visual-perceptual demands on TMT by subtracting completion time for TMT Part A from completion time for Part B (TMT B - A). TMT Part B-A provides a relatively purer measure of executive functioning. It has a timed scale from 0 sec (min) to 300 secs (max). Along this scale, a lower score is better.
Time Frame: 12 months
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Candesartan | Lisinopril
Number analyzed (Participants) | 87 | 89
seconds | 87.23 (5.46) | 111.37 (5.89)
Statistical Analysis 1: Comparison: Candesartan vs Lisinopril; All analyses were conducted using the intention-to-treat principle. Results are provided as adjusted least-square means with SE and effect size (ES) estimates (calculated from mixed model with repeated measures (MMRM) as the adjusted difference in cognitive change between the 2 groups over the study period); Test type: Superiority; Treatment effect size = -13.6, 95% CI 2-sided [-23.6 to -3.7] — effect size p-value = 0.008

2. Primary Outcome: NINDS-initiated EXecutive Abilities: Measures and Instruments for Neurobehavioral Evaluation and Research or "EXAMINER" Tool Box.
Description: EXecutive Abilities: Measures and Instruments for Neurobehavioral Evaluation and Research or "EXAMINER" tool box. This test batteryThe battery includes 11 tasks that generate 15 primary variables. Within this set, the EXAMINER includes: working memory, inhibition, set shifting, and fluency. The parts of EXAMINER that were used for this study include: Flanker task (inhibition) which involves responding to a central stimulus while ignoring flanking stimuli that are either compatible or incompatible with the central stimulus; Set-shifting, a measure of mental flexibility; Spatial 1-Back test assesses spatial working memory; Dot Counting test assesses verbal working memory; Verbal Fluency tested using a List Generation test which require the participant to generate words beginning with a specific letter, and category fluency in which the participant generates words from a specified category (e.g., animals, fruits). Higher are reflective of better executive function (-1 to +1)
Time Frame: 12 months
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Candesartan | Lisinopril
Number analyzed (Participants) | 87 | 89
units on a scale | 0.07 (0.07) | 0.25 (0.07)

3. Secondary Outcome: Memory
Description: To assess episodic memory, the Hopkins Verbal Learning Test-Revised (HVLT-R) will be used. The retention (%) score is calculated by dividing the delayed recall trial by the higher of 3 learning trials. Each trial scores 0 (min) to 12 (max). The HVLT-R retention score is a percentage, and a higher percentage represents a better outcome.
Time Frame: 12 months
Measure: Least Squares Mean (Standard Error); unit: percentage of retention
Arm/Group | Candesartan | Lisinopril
Number analyzed (Participants) | 87 | 89
percentage of retention | 82.71 (3.26) | 79.47 (3.39)

4. Secondary Outcome: Language
Description: This will be measured using the Boston Naming Test. BNT is a neuropsychological test used to assess visual confrontation naming and language performance in participants with cognitive decline. Its short 15-item version consists of drawings of objects ranging from common objects to less familiar objects. Scale: 0 (min score) to 15 (max score). For this test, a higher score/response represents a better outcome.
Time Frame: 12 months
Measure: Least Squares Mean (Standard Error); unit: number of correct responses
Arm/Group | Candesartan | Lisinopril
Number analyzed (Participants) | 87 | 89
number of correct responses | 13.42 (0.18) | 13.84 (0.18)

5. Secondary Outcome: Attention Measured Using Digit Span Backward
Description: The Digit Span test is a subtest of both the Wechsler Adult Intelligence Scale (WAIS) and the Wechsler Memory Scales (WMS). For the digit span backwards, subjects are read a sequence of numbers and asked to repeat the same sequence back to the examiner in reverse order (backward span). Backward span is an executive task particularly dependent on working memory. The Digit Span backward is scored for backwards performance. Scale: 0 (minimum) to 16 (maximum). A higher score represents a better outcome.
Time Frame: 12 months
Measure: Least Squares Mean (Standard Error); unit: Number of correct responses
Arm/Group | Candesartan | Lisinopril
Number analyzed (Participants) | 87 | 89
Number of correct responses | 5.14 (0.25) | 5.16 (0.26)

6. Secondary Outcome: White Matter Lesion Volume
Description: White Matter Lesion volume: high-resolution anatomical images are acquired for the measurement of microvascular disease. WMH volumes will be obtained from Fluid attenuated inversion recovery (FLAIR) imaging sequence and reported as total volume (in mm3). Higher values means greater WMH
Time Frame: 12 months
Population: Of 176 randomized participants, 27 did not complete an MRI scan at baseline (15 had metal implants with either pacemaker, stent, or inferior vena cava filter and 12 were claustrophobic). Of 141 participants who returned for their 12-month visit, an additional 8 participants refused to have a follow-up MRI. The final sample with both baseline and 12-month MRI was 104 participants (73.8%), including 51 participants in the candesartan group and 53 participants in the lisinopril group.
Measure: Least Squares Mean (Standard Error); unit: mm^3
Arm/Group | Candesartan | Lisinopril
Number analyzed (Participants) | 51 | 53
mm^3 | 2.68 (1.23) | 5.73 (1.22)

7. Secondary Outcome: Cerebral Perfusion
Description: ASL-MRI: Arterial Spin Labeling (ASL) MRI is non-invasive measure of perfusion that does not require contrast, and allows multiple brain regions mapping of perfusion and reserve. ASL-MRI provides measures of cerebral blood flow (CBF). Higher values indicates higher CBF.
Time Frame: 12 months
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: ml/100g/min
Arm/Group | Candesartan | Lisinopril
Number analyzed (Participants) | 51 | 53
ml/100g/min | 45.48 (1.47) | 47.65 (1.08)

8. Secondary Outcome: Attention Measured Using Digit Span Forward
Description: This will be measured using Digit Span Forward. The Digit Span test is a subtest of both the Wechsler Adult Intelligence Scale (WAIS) and the Wechsler Memory Scales (WMS). For the digit span forward, subjects are read a sequence of numbers and asked to repeat the same sequence back to the examiner in the correct order (forward span). Forward span captures attention efficiency and capacity. The Digit Span forward is scored for forwards performance. Scale: 0 (minimum) to 16 (maximum). A higher score represents a better outcome.
Time Frame: 12 months
Measure: Least Squares Mean (Standard Error); unit: Number of correct responses
Arm/Group | Candesartan | Lisinopril
Number analyzed (Participants) | 87 | 89
Number of correct responses | 9.67 (0.61) | 8.93 (0.66)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Candesartan | Lisinopril
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/89
Serious Adverse Events (participants affected / at risk) | 0/87 | 0/89
Other Adverse Events (participants affected / at risk) | 87/87 | 89/89
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Candesartan (N=87) | Lisinopril (N=89)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 24 (24)
Headache (General disorders) | 18 (18) | 22 (22)
Dizziness (General disorders) | 15 (15) | 14 (14)
Edema (General disorders) | 13 (13) | 12 (12)
General Pain (General disorders) | 7 (7) | 9 (9)
Fatigue (General disorders) | 9 (9) | 7 (7)
Nasal/sinus drainage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6)
Palpitation (Cardiac disorders) | 4 (4) | 4 (4)
Frequent urination (Renal and urinary disorders) | 4 (4) | 3 (3)
Leg Cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Insomnia (General disorders) | 0 (0) | 2 (2)
Runny nose (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Unusual bleeding or bruising (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Falling (General disorders) | 3 (3) | 1 (1)
Dry mouth (General disorders) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Loss of appetite (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Severe elevation in systolic BP >200 mmHg (Vascular disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 8 (8) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sweating (General disorders) | 0 (0) | 1 (1)
Fainting (General disorders) | 1 (1) | 0 (0)
Worsening renal function (serum creatinine >2.5) (Renal and urinary disorders) | 1 (1) | 0 (0)
Low potassium (<3.0) (Metabolism and nutrition disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
A limitation of this study is its 1-year study period. Additional limitations include the relatively small sample size, which limited our power to correct for multiple comparisons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2017-10-12): https://cdn.clinicaltrials.gov/large-docs/64/NCT01984164/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2015-02-05): https://cdn.clinicaltrials.gov/large-docs/64/NCT01984164/Prot_SAP_001.pdf